CLINICAL TRIAL: NCT05152810
Title: Efficacy of Transcranial Magnetic Stimulation (TMS) in Smoking Cessation, Combining Withdrawal Stimulations Followed by Maintenance Stimulations to Prevent Relapse: a Single-center, Randomized, Controlled, Blinded Pilot Study
Brief Title: Effectiveness of Transcranial Magnetic Stimulation (TMS) in Smoking Cessation, Combining Withdrawal Stimulation Followed by Maintenance Stimulation to Prevent Relapse
Acronym: TABACSTIM 3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TROJAK 2021
Record Dates: First submitted 2021-11-24; First posted 2021-12-10 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Transcranial Magnetic Stimulation (Experimental)
  Interventions: Other: Transcranial Magnetic Stimulation sessions; Other: Evaluations
- Transcranial magnetic resonance imaging placebo (Placebo Comparator)
  Interventions: Other: Transcranial Magnetic Stimulation sessions; Other: Evaluations

INTERVENTIONS:
Other: Transcranial Magnetic Stimulation sessions — * 10 sessions daily from Monday to Friday (2 sessions/day, 15 minutes apart) during the 1st week = attack phase
  * 2 weekly maintenance sessions the following week (S2), then 1 weekly maintenance session the following 4 weeks (S3, S4, S5 and S6) = maintenance phase
Other: Evaluations — Before the first stimulation session, just after the 10th session, at 6 weeks, at 12 weeks and at 24 weeks.
  The assessment included the collection of AEs/EIGs, the TAC, the VAS on "desire to smoke", the TCQ, the QSU, BDI-II (except at S1), the CO tester, GoNoGo, the PQI and the ISI.

SUMMARY:
Smoking cessation is a public health priority. Tobacco is directly responsible for 75,000 deaths per year in France. Without help, less than 5% of smokers are still abstinent after 12 months of smoking cessation. The use of nicotine replacement therapy only increases the chances of successful smoking cessation by 2-3%.

Brain imaging research shows that the dorsolateral prefrontal cortex (DLPC) is involved in tobacco addiction. Disorders induced in the DLPC cause an irrepressible urge to smoke (craving) and largely explain relapse during smoking cessation.

Transcranial Magnetic Stimulation (TMS) could be a promising tool in the quest for an effective approach to smoking cessation. This technique is used for direct stimulation of the DLPC via a magnetic coil in order to reduce the cortical activity of the DLPC and thus to reduce cravings.

A first randomized controlled study using TMS was conducted at the University Hospital of Dijon in highly addicted smokers who had failed to quit with the usual withdrawal strategies. In this study, entitled Tabacstim 1, we found that the combination of nicotine substitutes (to reduce physical withdrawal symptoms) with 10 "attack" sessions of TMS (to reduce cravings) increased the rate of abstinence during the first 2 weeks of withdrawal (% abstinence = 88. However, in this study, the therapeutic effect of the nicotine-SMT combination was not prolonged once the stimuli were stopped. At 6 and 12 weeks from the start of withdrawal, abstinence rates in the active SMT and placebo SMT groups were no longer significantly different.

We therefore initiated a new study, entitled Tabacstim 2, to add maintenance brain stimulation to the Tabacstim 1 protocol after the "attack" sessions (this therapeutic scheme is classically used in the treatment of depression with TMS). This study started in July 2020 and will end very soon (71 inclusions completed out of the 78 expected).

In both Tabacstim 1 and Tabacstim 2, the stimulations are delivered at low frequency (1 Hz) on the right DLPC. However, a recently published meta-analysis shows that, in addictions, stimulations delivered at a high frequency (10 Hz) on the left DLPC appear to be more effective in reducing craving. But above all, another meta-analysis carried out by our team (in progress of publication), finds that excitatory stimulations (such as 10 Hz rTMS) on the left DLPC are very effective in maintaining smoking abstinence in the medium term (3 and 6 months), which does not seem to be the case for inhibitory stimulations (such as 1 Hz rTMS).

We therefore wish to carry out the Tabacstim 3 study, which only differs from Tabacstim 2 in two stimulation parameters: 10 Hz stimulations on the left DLPC instead of 1 Hz stimulations on the right DLPC. We therefore propose in Tabacstim 3 to use excitatory stimulations on the left instead of inhibitory stimulations on the right.

Tabacstim 3 could be more effective for prolonged smoking cessation than the 2 previous protocols.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has given oral consent
* Adult patient
* Patient who wants to quit smoking
* Patient with a smoking disorder (DSM-5 criteria)
* Patient with at least 1 previous failed smoking cessation treatment with recommended medications (nicotine, vareniciline, or bupropion)

Exclusion Criteria:

* Patient not affiliated to the national health insurance system
* Patient subject to a measure of legal protection (curatorship, guardianship)
* Pregnant or breast-feeding woman
* Patient of childbearing age with a positive pregnancy test at inclusion
* Patients of legal age who are unable to express their consent
* Patient abstinent in the previous 3 months
* Patient with a substance use disorder (DSM-5 criteria)
* Patient with a contraindication to TMS: personal history of seizure, pacemaker, neurosurgical clips, carotid or aortic clips, heart valves, hearing aids, ventricular shunt valves, sutures with wires or staples, foreign bodies in the eye, shrapnel, other prosthesis or cephalic ferromagnetic material
* Patient employed in the addictology department of the CHU of Dijon (department of the principal investigator)
* Patient with severe depression, defined by a score greater than or equal to 24 on the Hamilton Depression Rating Scale (HDRS)
* Patient having had a recent change (< 1 month) in the prescription of a psychotropic treatment
* Patients with severe and/or chronic psychiatric disorders, including schizophrenia, paranoia, and bipolar disorder types I and II
* Patients with severe heart, kidney, liver or lung failure or other conditions that could compromise the patient's participation in the study in the opinion of the physician
* Patient concurrently participating in another therapeutic trial
* Patient who has already participated in a transcranial magnetic stimulation session

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-01-06 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Continuous Abstinence Rate | within 6 weeks of starting to quit smoking
  Continuous Abstinence Rate is defined according to Russell criteria as the proportion of patients reporting <5 cigarettes smoked since the 2nd week after the date of randomization (1 TMS session) AND biochemically validated by an expired carbon monoxide level of less than 10 ppm at follow-up and not contradicted by a previous self-report or validation result.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France